CLINICAL TRIAL: NCT04527445
Title: Reduction in Fluoroscopy Radiation Exposure During Lead Implantation for Sacral Neuromodulation: A Randomized Prospective Study
Brief Title: Fluoroscopy Radiation Reduction During Sacral Neuromodulation Lead Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5200182
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Radiation Exposure; Overactive Bladder; Urge Incontinence; Urgency-frequency Syndrome
Keywords: Sacral Neuromodulation; Fluoroscopy
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Masking Description: Subjects notified of the arm after the procedure is performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Radiation Fluoroscopy (Experimental): Reduced radiation fluoroscopy technique is performed by the C-arm set at 1 pulses-per-second and reduction of current.
  Interventions: Procedure: Reduced radiation fluoroscopy
- Conventional Fluoroscopy (Active Comparator): The standard of care is the conventional fluoroscopy, the C-arm is set at 30 pulses-per-second and the current set as the default.
  Interventions: Procedure: Conventional fluoroscopy

INTERVENTIONS:
Procedure: Reduced radiation fluoroscopy — See previous information about each arm
  Arms: Reduced Radiation Fluoroscopy
Procedure: Conventional fluoroscopy — See previous information about each arm
  Arms: Conventional Fluoroscopy

SUMMARY:
Fluoroscopy is performed when placing a lead during a sacral neuromodulation procedure. During lead placement, subjects will receive either conventional or experimental fluoroscopic settings. The radiation exposure will be compared between the two groups.

DETAILED DESCRIPTION:
Patients scheduled for lead implantation during sacral neuromodulation in the operating room and consent will be included in this study. Placement of the lead in the operating room with fluoroscopy is the standard of care in this procedure. Fluoroscopy is performed with a C-arm and there are settings that change the radiation exposure. Patients scheduled to undergo lead placement will be randomized to: a) the investigational (reduced radiation with fluoroscopic settings) or b. the control (conventional fluoroscopy).

The surgeon can change fluoroscopy radiation exposure by changing C-arm settings from the reduced radiation to conventional fluoroscopic options. During the surgery, the surgeon may change the settings from reduced radiation (intervention) to conventional fluoroscopy (control) to safely place lead. The surgeon will use their judgment to optimally place lead and maintain safety during placement. Any deviation from randomization will be recorded.

The intervention arm is defined: Reduced radiation fluoroscopy technique is performed by the C-arm set at 1 pulses-per-second and reduction of current.

The control arm is defined: The standard of care in the conventional fluoroscopy, the C-arm is set at 30 pulses-per-second and the current set at the default.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lead implantation for sacral neuromodulation that have overactive bladder as defined by urinary urgency, frequency, nocturia with or without urgency incontinence.

Exclusion Criteria:

* neurogenic bladder, BMI >40, or peripheral neuropathy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radiation Exposure | At time of procedure
  measure radiation exposure, milligray (mGy)

SECONDARY OUTCOMES:
Optimal lead placement | At time of procedure
  based on intraoperative motor response
Voiding log (Bladder Record) | 3 months after surgery
  Clinical Outcome
Clinical Outcome assessed by validated questionnaire | 3 months after surgery
Inoperative complications | At time of procedure
  surgery complication
Operative times | At time of procedure
  minutes

CONTACTS AND LOCATIONS:
Overall Officials: Forrest Jellison, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No